CLINICAL TRIAL: NCT05901532
Title: Nasal Irrigation With Chinese Herbal Medicine as an Adjunctive Treatment in Allergic Rhinitis: Phase 2 Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Nasal Irrigation With Chinese Herbal Medicine as an Adjunctive Treatment in Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF19289A
Record Dates: First submitted 2023-05-12; First posted 2023-06-13 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-06

CONDITIONS: Rhinitis, Allergic; Nasal Lavage; Medicine, Chinese Traditional
Keywords: Rhinitis, Allergic; Nasal Lavage; Medicine, Chinese Traditional
MeSH Terms: conditions — Rhinitis, Allergic | interventions — isoborneol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese herbal medicine (Experimental): The bilateral nasal cavity was irrigated with a bottle of NeilMed containing 1 gram of Szechwan Lovage Rhizome, 1 gram of Biod Magnolia Bud, 0.5 gram of Taiwan Angelica Root, 0.5 gram of Wild Mint Herb, 1.5 gram of Baikal Skullcap Root, and 0.5 gram of Borneol dissolved in 240 ml of warm normal saline once a day.
  Interventions: Drug: Szechwan Lovage Rhizome, Biod Magnolia Bud, Taiwan Angelica Root, Wild Mint Herb, Baikal Skullcap Root, and Borneol
- Placebo (Placebo Comparator): The bilateral nasal cavity was irrigated with a bottle of NeilMed containing edible caramel dissolved in 240 ml of warm normal saline once a day.
  Interventions: Drug: edible caramel

INTERVENTIONS:
Drug: Szechwan Lovage Rhizome, Biod Magnolia Bud, Taiwan Angelica Root, Wild Mint Herb, Baikal Skullcap Root, and Borneol — The bilateral nasal cavity was irrigated with a plastic bottle containing 1 gram of Szechwan Lovage Rhizome, 1 gram of Biod Magnolia Bud, 0.5 gram of Taiwan Angelica Root, 0.5 gram of Wild Mint Herb, 1.5 gram of Baikal Skullcap Root, and 0.5 gram of Borneol dissolved in 240 ml of warm normal saline once a day for 2 months.
  Arms: Chinese herbal medicine
Drug: edible caramel — The bilateral nasal cavity was irrigated with a plastic bottle containing edible caramel dissolved in 240 ml of warm normal saline once a day for 2 months.
  Arms: Placebo

SUMMARY:
In allergic rhinitis patients with severe symptoms, control of severe allergic reactions is limited with saline nasal irrigation. Therefore, there have been several attempts to use saline nasal irrigation in combination with other treatments to treat allergic rhinitis. This study tries to explore the effect of nasal irrigation with Chinese herbal medicines on allergic rhinitis.

DETAILED DESCRIPTION:
In this study, patients with allergic rhinitis over 20 years old were collected from the clinics of Otolaryngology and Traditional Chinese Medicine clinics. The subjects were randomly divided into two groups. They used the devices of NeiMed sinus rinse to irrigate the nose with 240 cc of Chinese herbal medicine solution or placebo each morning and evening for 2 months. Subjects in both groups filled questionnaires, and received acoustic rhinometry, rhinomanometry, and eustachian tube function tests before and after nasal irrigation. This study tries to explore the effect of nasal irrigation with Chinese herbal medicines on allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis patients diagnosed based on the history and allergen test

Exclusion Criteria:

* Those younger than 20 years old, Immunocompromised patients Pregnant women or breastfeeding women Those with a history of allergy to traditional Chinese medicine Those with liver and kidney insufficiency Those who cannot cooperate with nasal irrigation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change of rhinitis symptom score | Evaluated baseline and 2-month nasal lavage
  The effect of rhinorrhea, sneezing, nasal obstruction and itching on life quality was measuring by scores. Score 0 means no symptom, score 1 means symptomatic but not annoying, score 2 means troublesome symptoms and affecting part of daily activity or sleep and score 3 means annoying symptoms and affecting most daily activity or sleep.
Self-reported adverse events | Through study completion, an average of 2 months
  Any adverse events occurring during the study period

SECONDARY OUTCOMES:
Change of swollen degree of inferior turbinates | Evaluated baseline and 2-month nasal lavage
  The swollen degree of inferior turbinates was measuring by scores. Score 0 means inferior turbinates occupying less than 25% of nasal cavity, score 1 means inferior turbinates occupying 26 to 50 of nasal cavity, score 2 means inferior turbinates occupying 51 to 75 of nasal cavity and score 3 means inferior turbinates occupying more than 75% of nasal cavity.
Change of the second minimal cross-sectional area of the nasal cavity | Measured baseline and 2-month nasal lavage
  The second minimal cross-sectional area of the nasal cavity was measured by acoustic rhinometry.
Change of total inspiratory resistance | Measured baseline and 2-month nasal lavage
  Total inspiratory resistance was measured by rhinomanometry.
Change of score measured by Eustachian Tube Dysfunction Patient Questionnaire | Evaluated baseline and 2-month nasal lavage
  Using a 7-item Eustachian Tube Dysfunction Patient Questionnaire to evaluate Eustachian Tube function
Change of Eustachian Tube function test | Evaluated baseline and 2-month nasal lavage
  Performing a Eustachian Tube Function Test to evaluate Eustachian Tube function

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Rong-San Jiang, Taichung, Taiwan